CLINICAL TRIAL: NCT03372161
Title: Corticosteroid Lumbar Epidural Analgesia for Radiculopathy (C.L.E.A.R.)
Brief Title: Corticosteroid Lumbar Epidural Analgesia for Radiculopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other); Semnur Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP-102-02
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Results first posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-08

CONDITIONS: Lumbosacral Radicular Pain
Keywords: lumbosacral radicular pain; sciatica; leg pain
MeSH Terms: conditions — Sciatica

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SP-102 (Experimental): SP-102
  Interventions: Drug: SP-102
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-102 — injection
  Arms: SP-102
Drug: Placebo — injection
  Arms: Placebo

SUMMARY:
This is a research study of SP-102, an experimental medication designed to relieve pain in patients with a specific type of leg pain. The medication is given once by your healthcare professional, with a possibility of a second injection as early as about 1 month after the first treatment.

The purpose of the study is to measure how well a single injection of the experimental medication, SP-102, relieves pain. The study will also investigate the side effects of SP-102.

ELIGIBILITY:
Main Inclusion Criteria:

* Able and willing to read, write, and understand the English language and provide English language written informed consent prior to beginning any study procedures.
* Age 18 to 70 years (inclusive) at the Screening Visit.
* A diagnosis of lumbosacral radicular pain (sciatica).
* Agrees to follow study-specific medication requirements.
* If sexually active and a female of child-bearing potential or a male capable of bearing a child, agrees to use an effective method of birth control during the study.
* Has reviewed all study specific materials and has, in the opinion of the Investigator, the abilities to understand and appropriately complete all study procedures.

Main Exclusion Criteria:

* Has radiologic evidence of a condition that would compromise study outcomes.
* Has ever had lumbosacral back surgery or plans to undergo spine surgical intervention while in the study.
* Has been diagnosed with insulin dependent diabetes mellitus.
* Presence of any other disorder, condition or circumstance (including secondary gain) that, in the opinion of the Investigator, has the potential to prevent study completion and/or to have a confounding effect on outcome assessments.
* Use of any investigational drug and/or device within 30 days, or is scheduled to receive an investigational drug other than blinded study drug during this study.
* Has a body mass index ≥40 kg/m2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2022-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Lissin, MD, Study Director — Scilex Pharmaceuticals, Inc.
Locations (37):
- United States (37):
  - Semnur Research Site 75, Mobile, Alabama
  - Semnur Research Site 52, Phoenix, Arizona
  - Semnur Research Site 58, Tempe, Arizona
  - Semnur Research Site 18, La Jolla, California
  - Semnur Research Site 47, Laguna Woods, California
  - Semnur Research Site 70, Los Gatos, California
  - Semnur Research Site 56, Fernandina Beach, Florida
  - Semnur Research Site 81, Jacksonville, Florida
  - Semnur Research Site 49, St. Petersburg, Florida
  - Semnur Research Site 13, Tampa, Florida
  - Semnur Research Site 61, Tampa, Florida
  - Semnur Research Site 53, Winter Park, Florida
  - Semnur Research Site 28, Marietta, Georgia
  - Semnur Research Site 64, Marietta, Georgia
  - Semnur Research Site 10, Newnan, Georgia
  - Semnur Research Site 38, Boise, Idaho
  - Semnur Research Site 40, Bloomington, Illinois
  - Semnur Research Site 63, Chicago, Illinois
  - Semnur Research Site 12, Chicago, Illinois
  - Semnur Research Site 19, Chicago, Illinois
  - Semnur Reseach Site 62, Overland Park, Kansas
  - Semnur Research Site 51, Burlington, Massachusetts
  - Semnur Research Site 65, Omaha, Nebraska
  - Semnur Research Site 60, Las Vegas, Nevada
  - Semnur Research Site 30, Shrewsbury, New Jersey
  - Semnur Research Site 11, Durham, North Carolina
  - Semnur Research Site 20, Winston-Salem, North Carolina
  - Semnur Research Site 46, Cleveland, Ohio
  - Semnur Research Site 43, Cuyahoga Falls, Ohio
  - Semnur Research Site 36, Oklahoma City, Oklahoma
  - Semnur Research Site 48, Charleston, South Carolina
  - Semnur Research Site 77, Greenville, South Carolina
  - Semnur Research Site 15, Houston, Texas
  - Semnur Research Site 54, Plano, Texas
  - Semnur Research Site 35, Tyler, Texas
  - Semnur Research Site 59, Draper, Utah
  - Semnur Research Site 42, Greenfield, Wisconsin

REFERENCES:
- [Derived] Miller A, Candido KD, Knezevic NN, Rivera J, Lunseth P, Levinson DJ, Formoso F, Solanki D, Tavel E, Krull A, Radnovich R, Burkhead D, Souza D, Helm S, Katz N, Dworkin RH, Cohen SP, Rathmell JP, Buvanendran A, Levin J, Stannard E, Ambrose C, Jaros M, Vought K, Lissin D. A randomized, placebo-controlled trial of long-acting dexamethasone viscous gel delivered by transforaminal injection for lumbosacral radicular pain. Pain. 2024 Dec 1;165(12):2762-2773. doi: 10.1097/j.pain.0000000000003287. Epub 2024 Jun 14. PMID 38875121

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SP-102 | Placebo
Started | 202 | 199
Completed | 193 | 192
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SP-102 | Placebo | Total
Number analyzed (Participants) | 202 | 199 | 401
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (9.83) | 51.7 (10.36) | 51.4 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 122 | 238
  Male | 86 | 77 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 35 | 69
  Not Hispanic or Latino | 168 | 164 | 332
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 33 | 70
  White | 160 | 162 | 322
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Day 1) to Week 4 in the Mean Numeric Pain Rating Scale (NPRS) Average Pain Score in the Affected Leg
Description: The NPRS is an 11-point scale (0 to 10-point scale where 0 was no pain and 10 was worst pain imaginable) that allowed the subject to rate the severity of their pain intensity at various points in time.
Time Frame: Baseline, 4 Weeks
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | SP-102 | Placebo
Number analyzed (Participants) | 148 | 184
Change in score on a scale from baseline | -2.34 (1.842) | -1.16 (1.723)

2. Secondary Outcome: Mean Change From Baseline (Day 1) to Week 4 in the Oswestry Disability Index Score (ODI)
Description: The ODI is the gold standard for measuring degree of disability and estimating quality of life in a person with low back pain. The ODI is a questionnaire completed by the subject that assesses10 topics: intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each question was scored on a scale of 0-5 with 0 indicating the least amount of disability and 5 indicating the most severe disability. The scores for all questions answered were summed, then multiplied by 2 to obtain the index (range 0 to 100). Zero was equated with no disability and 100 was the maximum disability possible.
Time Frame: Baseline, 4 Weeks
Measure: Mean (Standard Deviation); unit: Change in score on a scale from baseline
Arm/Group | SP-102 | Placebo
Number analyzed (Participants) | 147 | 177
Change in score on a scale from baseline | -10.89 (14.906) | -4.76 (12.896)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | SP-102 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/202 | 1/199
Serious Adverse Events (participants affected / at risk) | 0/202 | 2/199
Other Adverse Events (participants affected / at risk) | 60/202 | 42/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SP-102 (N=202) | Placebo (N=199)
Cardiac arrest (Cardiac disorders) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SP-102 (N=202) | Placebo (N=199)
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Toothache (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 1
Gait disturbance (General disorders) | 1 | 0
Injection site pain (General disorders) | 4 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 2
COVID-19 (Infections and infestations) | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Dacryocystitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 4 | 0
Tooth abscess (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 3
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 2 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Blood pressure increased (Investigations) | 2 | 0
Cardiac murmur (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Burning sensation (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Formication (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 13 | 11
Hypoaesthesia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 3 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Radicular pain (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Accelerated hypertension (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has the right to first publication of the results of the study. Following the first publication, PIs may publish study data or results; however, the proposed publication must be submitted to the Sponsor for review and approval in writing at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study Data.

DOCUMENTS (2):
  • Study Protocol (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT03372161/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT03372161/SAP_001.pdf